CLINICAL TRIAL: NCT04460898
Title: Real-World Treatment Patterns and Outcomes in Postmenopausal, Hormone-Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative, Metastatic Breast Cancer Patients Treated With Palbociclib Plus an Letrozole as Initial Endocrine Therapy at Community Oncology Practices in the U.S.
Brief Title: RW Treatment Patterns and Outcomes in Postmenopausal HR+/HER2- mBC Patients Treated With Palbociclib Plus Letrozole as Initial Endocrine Therapy at Community Oncology Practices in the U.S.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481123
Record Dates: First submitted 2020-07-06; First posted 2020-07-08 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Breast Cancer Patients: HR+/HER2- metastatic breast cancer patients in the US.

SUMMARY:
This is a retrospective, observational study that will document treatment patterns and clinical outcomes of postmenopausal patients diagnosed with HR+/HER2- mBC who received Palbociclib plus Letrozole as initial endocrine-based therapy in US community oncology network settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

  1. Diagnosed with locoregional recurrent or metastatic female breast cancer.
  2. Pathologically confirmed HR-positive/HER2-negative diagnosis.
  3. Received treatment with palbociclib in combination with letrozole as initial endocrine-based therapy for advanced/metastatic breast cancer:

     1. Initiated treatment with palbociclib at least 3 months following the provider's first use of palbociclib following its FDA approval.
     2. At least 1 month of follow-up (at least one visit with the provider) after initiation of palbociclib.
  4. Postmenopausal (or receiving surgical or medical treatment to induce menopause) at the time of initiation of palbociclib.
  5. ≥18 year old at initiation of palbociclib.

     Exclusion Criteria:
* No exclusion criteria will be imposed for the selection of patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients aged 18 years and older, diagnosed with HR+/HER2- mBC and received treatment with Palbociclib in combination with letrozole as initial endocrine-therapy for advanced/metastatic breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer United States, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481123

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data of metastatic breast cancer participants who received palbociclib and letrozole (LET) as initial endocrine therapy on or after 03 February 2015 up to Feb 11, 2019 (approximately 4 years) at community oncology practices in the U.S. as per FDA approval labels, were observed retrospectively. Data from medical records of eligible participants were collected by their treating physician. Data were identified and evaluated for 5.7 months approximately in this observational study.
Groups:
- Palbociclib + LET: Participants received palbociclib along with LET as initial endocrine-based therapy for advanced and metastatic breast cancer per FDA approval labels as part of their routine treatment. Data were retrieved and observed retrospectively for a period of 5.7 months approximately in this study.
Period: Overall Study
Arm/Group | Palbociclib + LET
Started | 195
Completed | 195
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who after clinical and analytical quality control assessment were retained for analysis in the study.
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.92 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 170
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 33
  White | 145
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to Year of Initial Diagnosis of Breast Cancer
Description: Number of participants according to their year of initial diagnosis of breast cancer were reported.
Time Frame: Baseline during data identification period of approximately 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: FAS included all participants who after clinical and analytical quality control assessment were retained for analysis in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Participants
  Prior to 2011 | 27
  Jan 2011 to Dec 2014 | 28
  Jan 2015 to Dec 2018 | 139
  Jan 2019 | 1

2. Primary Outcome: Number of Participants With American Joint Committee on Cancer (AJCC) Stage Status
Description: AJCC stages included: stage l (T1N0M0), stage IIA (T0N1M0, T1N1M0, T2N0M0), stage IIB (T2N1M0, T3N0M0), stage IIIA (T0N2M0, T1N2M0, T2N3M0, T3N1 or N2M0), stage IIIB (T4 any NM0, any TN3M0), stage IIIC (any TN3M0), stage IV (any T any NM1), and unknown. T0 = early form of tumor, T1 = less than (<) 2 centimeter (cm), T2 =2-5 cm, T3 = greater than (>) 2 cm, T4 = large sized, N0 = not spread to lymph node (LN), N1 = spread to LN 1 to 3, N2= spread to LN 4 to 9, N3 = spread >10 axillary LN, M0 = no metastasis, M1= metastasis.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Participants
  Stage I | 15
  Stage IIA | 16
  Stage IIB | 17
  Stage IIIA | 11
  Stage IIIB | 4
  Stage IIIC | 3
  Stage IV | 128
  Unknown | 1

3. Primary Outcome: Number of Participants With Node Status
Description: In this outcome measure, number of participants with node status ranging from N0 to Nx were recorded and reported. N0= No regional lymph node involvement (no cancer found in the lymph nodes), N1-N3= involvement of regional lymph nodes (number and/or extent of spread), and Nx = regional lymph nodes cannot be evaluated. N2 included N2A, and N2B stages; N3 included N3A, N3B, and N3C stages.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Participants
  N0 | 44
  N1 | 44
  N2A | 14
  N2B | 10
  N3A | 6
  N3B | 4
  N3C | 7
  Nx | 66

4. Primary Outcome: Number of Participants With Menopausal Status
Description: In this outcome measure, number of participants with menopausal status were recorded and reported. Menopausal status included pre-menopausal, peri-menopausal and post-menopausal.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Participants
  Pre-menopausal | 7
  Peri-menopausal | 5
  Post-menopausal | 183

5. Primary Outcome: Number of Participants With Type of Metastatic Disease
Description: In this outcome measure, number of participants with de novo metastatic and recurrent types of metastatic disease were recorded and reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Participants
  De novo metastatic | 128
  Recurrent metastatic | 67

6. Primary Outcome: Number of Participants With Sites of Metastatic Disease
Description: Sites of metastatic disease included: locoregional site, adrenal gland, bone, brain, distant lymph nodes, gastrointestinal system, liver, lung, pleura, pericardial, and/or peritoneal cavity. A participant could have more than 1 metastatic site.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Participants
  Locoregional site | 8
  Adrenal gland | 12
  Bone | 141
  Brain | 2
  Distant lymph nodes | 47
  Gastrointestinal system | 1
  Liver | 24
  Lung | 69
  Pleura, pericardial, and/or peritoneal cavity | 8

7. Primary Outcome: Number of Participants With Total Number of Metastatic Sites
Description: In this outcome measure, number of participants with total number of metastatic sites ranging from 1 to >3 were recorded and reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Participants
  1 | 82
  2 | 78
  >3 | 35

8. Primary Outcome: Number of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG-PS) at the Time of Initiation of First-line Treatment
Description: In this outcome measure, number of participants with ECOG at the time of initiation of first-line treatment were included. ECOG scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature; 2= ambulatory and capable of all self-care, but unable to carry out any work activities, up and about >50 percent (%) of waking hours; 3=capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair.
Time Frame: Pre-dose on Day 1 of treatment during data identification period of approximately 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Participants
  ECOG Status: 0 | 68
  ECOG Status: 1 | 107
  ECOG Status: 2 | 17
  ECOG Status: 3 | 3
  ECOG Status: 4 | 0

9. Primary Outcome: Number of Participants With Comorbidities at the Time of Initiation of First-line Treatment
Description: In this outcome measure, number of participants with various comorbidities at the time of initiation of first-line treatment were recorded and reported. Comorbidities included acquired immune deficiency syndrome/human immune virus (AIDS/HIV), cardiovascular disease, cerebrovascular disease, chronic pulmonary disease, congestive heart failure, connective tissue disease, dementia, depression, diabetes with chronic complications, diabetes without chronic complications, hemiplegia or paraplegia, hypertension, liver disease - mild, moderate, or severe, myocardial infarction, other hematologic malignancy, other non-hematologic malignancy, peptic ulcer disease, peripheral vascular disease, renal disease, thromboembolic events (arterial or venous), and other. One participant could have more than 1 comorbidity. Data with "0" values has not been reported in this outcome measure.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Participants
  Cardiovascular disease | 25
  Cerebrovascular disease | 6
  Chronic pulmonary disease | 9
  Congestive heart failure | 7
  Connective tissue disease | 4
  Dementia | 3
  Depression | 22
  Diabetes with chronic complications | 4
  Diabetes without chronic complications | 26
  Hypertension | 109
  Liver disease - mild | 3
  Myocardial infarction | 2
  Peptic ulcer disease | 8
  Peripheral vascular disease | 1
  Renal disease | 5
  Thromboembolic events (arterial or venous) | 4
  Other | 10

10. Primary Outcome: Charlson Comorbidity Index (CCI) Score
Description: CCI based on various comorbid conditions including myocardial infarction, congestive heart failure, peripheral vascular disease, cerebrovascular disease, dementia, chronic pulmonary disease, rheumatologic disease, peptic ulcer disease, hemiplegia or paraplegia, renal disease, AIDS/HIV, diabetes with and without chronic complications, liver disease (mild, moderate, or severe) was reported. CCI score range was from 0 to 14, where 0= low comorbid condition and 14= high comorbid condition, higher scores indicated more comorbidity.
Time Frame: Day 1 of treatment during data identification period of approximately 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Units on a scale | 0.52 (0.93)

11. Primary Outcome: Number of Participants Who Received Chemotherapy (Neo/Adjuvant) and Hormonal Therapy
Description: In this outcome measure, number of participants who received neo/adjuvant chemotherapy and hormonal (endocrine) therapy were recorded and reported. Neo/Adjuvant chemotherapy and hormonal therapy were the treatments administered before primary cancer treatment to enhance the outcome of primary treatment. Participants reported in rows below are not mutually exclusive.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Participants
  Adjuvant chemotherapy | 31
  Adjuvant endocrine therapy | 51
  Both adjuvant chemotherapy/adjuvant endocrine therapy | 25

12. Primary Outcome: Duration of Adjuvant Therapy
Time Frame: as for outcome 1
Population: FAS included all participants who after clinical and analytical quality control assessment were retained for analysis in the study. Here 'Overall Number of Participants Analyzed' = number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 57
Months | 41.7 (28.16)

13. Primary Outcome: Time From Discontinuation of Adjuvant Therapy to Initiation of First-line Treatment
Description: In this outcome measure, time from discontinuation (in months) of adjuvant therapy up to the initiation of first-line treatment of palbociclib combination was recorded and reported.
Time Frame: as for outcome 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 57
Months | 39.32 (50.81)

14. Primary Outcome: Number of Participants With Different Initial Palbociclib Dose
Description: In this outcome measure, number of participants with different initial dose treatment patterns (125 milligram [mg]/day, 100 mg/day, and 75 mg/day) at palbociclib initiation were recorded and reported.
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 193
Participants
  125 mg/day | 166
  100 mg/day | 26
  75 mg/day | 1

15. Primary Outcome: Total Number of Treatment Cycles Received
Description: Total number of cycles of treatment was the mean number of cycles received by participants prior to the discontinuation of initial treatment of metastatic breast cancer.
Time Frame: From first-line treatment up to the discontinuation of initial treatment of metastatic breast cancer during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Cycles
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 193
Cycles | 13.73 (10.10)

16. Primary Outcome: Number of Participants With Dose Reductions
Description: In this outcome measure, number of participants whose dose was reduced from 125 mg/day to 100 mg/day or from 125 mg/day to 75 mg/day, or from 100 mg/day to 75 mg/day were recorded and reported.
Time Frame: From start to end of treatment during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 193
Participants | 33

17. Primary Outcome: Number of Participants With Increased Dose Patterns
Description: In this outcome measure, number of participants with increased dose patterns from 100 mg/day to 125 mg/day, 75 mg/day to 125 mg/day, and from 75 mg/day to 100 mg/day were recorded and reported.
Time Frame: as for outcome 16
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 193
Participants | 0

18. Primary Outcome: Number of Participants With Any Treatment Interruptions
Description: In this outcome measure, number of participants whose treatment was interrupted due to any reason (toxicity, no response, loss of response, disease progression (PD), prepare for alternative treatment strategy, participant choice or other) were recorded and reported.
Time Frame: as for outcome 16
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 193
Participants | 17

19. Primary Outcome: Frequency of CBC Testing During First Cycle of Treatment
Description: In this outcome measure, mean of number of complete blood count (CBC) testing was recorded during first cycle of first line (1L) treatment. 1 cycle was of 28 days.
Time Frame: During first cycle of first line treatment during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: CBC testing
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 192
CBC testing | 2.07 (1.06)

20. Primary Outcome: Frequency of Electrolyte Testing During First Cycle of First Line Treatment
Description: In this outcome measure, mean of number of electrolyte testing was recorded during first cycle of first line treatment. 1 cycle was of 28 days.
Time Frame: as for outcome 19
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Electrolyte testing
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 190
Electrolyte testing | 1.44 (0.89)

21. Primary Outcome: Frequency of Liver Function Testing During First Cycle of First Line Treatment
Description: In this outcome measure, mean of liver function testing was recorded during first cycle of first line treatment. 1 cycle was of 28 days.
Time Frame: as for outcome 19
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Liver function testing
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 191
Liver function testing | 1.37 (0.76)

22. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS) at Month 6
Description: PFS= time from 1L Palbociclib combination treatment initiation until clinician documented PD while on Palbociclib/death. Participants who discontinued 1L treatment due to toxicity, participant's choice/other reason were censored on date of discontinuation. PD=increase in visible disease &/or presence of any new lesion; included cases where clinician indicated PD. Percentage of participants who were progression-free & alive at 6 months following palbociclib initiation was calculated by Kaplan-Meier method. Event (PD/death) = any record of measurable increase in disease (size of lesion at initiation of palbociclib versus most recent scan), presence of new lesions (new sites based on most recent scan/biopsy), notation in participants electronic health record by treating physician that participant had progressed/recorded date of death. Participants were censored if they discontinued 1L treatment with palbociclib due to any reason other than PD/death (toxicity/participant request, etc).
Time Frame: Month 6 during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Percentage of participants | 92.7 [87.5 to 95.8]

23. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS) at Month 12
Description: as for outcome 22
Time Frame: Month 12 during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Percentage of participants | 75.5 [67.5 to 81.9]

24. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS) at Month 18
Description: as for outcome 22
Time Frame: Month 18 during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Percentage of participants | 51.6 [42.4 to 60.0]

25. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS) at Month 24
Description: as for outcome 22
Time Frame: Month 24 during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Percentage of participants | 42.0 [32.7 to 51.0]

26. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the interval from the initiation of first line palbociclib combination treatment until death. Participants who were alive at the time of data collection were censored on the last date of visit with their provider.
Time Frame: From initiation of treatment up to death during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Months | NA [41.9 to NA] — Median and upper limit for 95% CI could not be estimated because there were insufficient number of participants with event.

27. Primary Outcome: Percentage of Participants With Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants who achieved complete (where 'complete response' was recorded at any time on treatment) or partial response (where 'partial response' was recorded at any time on treatment), or stable disease at greater than equal to (>=) 24 weeks on palbociclib combination therapy. Stable disease was defined as no evidence of complete or partial response, and no progression on palbociclib therapy for 24 weeks or greater. Complete response: Complete resolution of all visible disease. Partial response: Partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease
Time Frame: From initiation of treatment up to CR and PR and SD during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Percentage of participants | 83.08

28. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved complete response (CR) or partial response (PR) on palbociclib combination therapy recorded from first dose of study treatment until disease progression due to any cause. Complete response: complete resolution of all visible disease. Partial response: partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease.
Time Frame: as for outcome 27
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 195
Percentage of participants | 65.13

29. Primary Outcome: Number of Participants With Stable Disease Lasting Greater Than (>) 24 Weeks
Description: Stable disease was defined as no evidence of complete or partial response, and no progression on palbociclib therapy for 24 weeks or greater. Complete response: Complete resolution of all visible disease. Partial response: Partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease.
Time Frame: From initiation of treatment up to end of treatment during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 162
Participants | 35

30. Primary Outcome: Number of Participants Who Received Drug Regimen Post Discontinuation of Initial Endocrine-Based Therapy
Description: In this outcome measure, number of participants who received drug regimen after discontinuation of initial endocrine-based therapy were recorded and reported.
Time Frame: Post discontinuation of initial endocrine-based therapy during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 76
Participants
  Chemotherapy | 44
  Endocrine therapy | 28
  Other therapy | 4

31. Primary Outcome: Duration of Discontinued Therapy
Description: Discontinuation referred to a treatment persistence terminal event other than regimen change or switch, disease progression, or death. Participants who had a termination of palbociclib for reasons other than regimen change or switch, disease progression, or death were recorded and reported as discontinued.
Time Frame: Up to 24 months after palbociclib treatment initiation during data identification of approximatively 4 years (from the data retrieved and observed retrospectively over a duration of 5.7 months)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Palbociclib + LET
Number analyzed (Participants) | 18
Months | 8.48 (2.54)

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not planned to be collected and evaluated during the study
Description: Due to non-interventional nature of the study, safety data was not collected. The study was a retrospective study of existing medical records, and focused on treatment patterns and effectiveness outcomes. There was no collection of adverse events in the study, so there is no report of adverse events in the results.
Arm/Group | Palbociclib + LET
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04460898/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04460898/SAP_001.pdf